CLINICAL TRIAL: NCT01258270
Title: Efficacy and Patient Satisfaction With AQUACEL® Ag Surgical Dressing Compared to Standard Surgical Dressing. A Prospective, Randomized Study in Primary Total Joint Arthroplasty.
Brief Title: Efficacy and Patient Satisfaction With AQUACEL® Ag Surgical Dressing Compared to Standard Surgical Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-10-01A
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2012-01

CONDITIONS: Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (AQUACEL® Ag Surgical Dressing (Active Comparator)
  Interventions: Procedure: Postop Dressing
- Standard island gauze and tape dressing (Active Comparator): A standard island dressing consists of adhesive tape and gauze.
  Interventions: Procedure: Postop Dressing

INTERVENTIONS:
Procedure: Postop Dressing — The AQUACEL® Ag Surgical Dressing is a silver impregnated, waterproof, adhesive dressing that sticks to the skin around the wound and blocks bacteria from the outside.
  Arms: (AQUACEL® Ag Surgical Dressing
Procedure: Postop Dressing — A standard island dressing consists of adhesive tape and gauze.
  Arms: Standard island gauze and tape dressing

SUMMARY:
The objective of this study is to determine the safety and effectiveness of the AQUACEL® Ag Surgical Dressing (treatment group) as compared to prepackaged island wound dressings consisting of traditional tape and gauze (control group) for total hip and total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting for primary total hip performed through a posterior or posterior-lateral surgical approach or primary total knee arthroplasty
2. Patients between the ages of 18 and 90
3. The subject is willing and able to understand, sign and date the study specific patient Informed Consent, to volunteer participation in the study
4. The subject is having surgery at a Carolinas HealthCare System facility
5. The subject is psychosocially, mentally and physically able to comply with the requirements of the study

Exclusion Criteria:

1. Patients presenting for revision total hip or total knee arthroplasty
2. Patients with topical hypersensitivity or allergy to any disposable components of the dressing system such as: ionic silver, polyurethane film
3. Any systemic or local active dermatological disease that might interfere with the evaluation of the surgical site such as eczema, psoriasis, skin cancer, scleroderma, chronic urticaria
4. Patients currently participating in another clinical trial that may affect your participation in this trial
5. Patients with insurance coverage not included in Gentiva list of payers
6. Patients residing outside of Gentiva's geographical coverage area
7. Patients having surgery at a NON-Carolinas HealthCare System facility

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative severe skin reactions (defined as blisters) around the surgical incision site | 4 weeks postop
  Wound checks will be performed during the postoperative period in the hospital followed by home healthcare providers. The final wound check will be performed by the surgeon at 4 weeks postoperatively.

SECONDARY OUTCOMES:
Patient pain and satisfaction (1-100 visual analog scale) | immediate postop, 5-7 days postop, 4 weeks postop

CONTACTS AND LOCATIONS:
Overall Officials: Bryan D Springer, MD, Principal Investigator — OrthoCarolina, PA
Locations (1):
- OrthoCarolina, PA, Charlotte, North Carolina, United States